CLINICAL TRIAL: NCT06068296
Title: Towards a Clinical Test Battery for the Assessment of Verbal Short-term Memory Abilities With Linguistic Variations in Patients With Poststroke Aphasia.
Brief Title: Short-term Memory Assessment in Patients With Poststroke Aphasia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: BC-08865
Record Dates: First submitted 2022-12-21; First posted 2023-10-05 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-09

CONDITIONS: Aphasia, Acquired; Short-Term Memory Impairment
Keywords: aphasia; short-term memory; assessment
MeSH Terms: conditions — Aphasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Short term memory assessment in patients with aphasia. (Other): Evaluation of short term memory in a patient population with poststroke aphasia using a dutch version of the Temple Assessment of Language and Verbal Short-Term memory in aphasia (TALSA).
  Interventions: Diagnostic Test: short term memory assessment; Diagnostic Test: Oxford cognitive screen; Diagnostic Test: Token Test
- short term memory assessment in healthy volunteers (Other): Evaluation of short term memory in healthy volunteers using a dutch version of the Temple Assessment of Language and Verbal Short-Term memory in aphasia (TALSA).
  Interventions: Diagnostic Test: short term memory assessment; Diagnostic Test: Montreal cognitive assessment

INTERVENTIONS:
Diagnostic Test: short term memory assessment — Aphasia group: The Dutch verbal STM assessment tool will be administered over a time span of maximum two consecutive days depending on how fatigued the patient is during testing.
  Healthy control group: the Dutch verbal STM assessment tool will be administered.
Diagnostic Test: Oxford cognitive screen — Evaluation of the cognitive abilities of the patients with aphasia.
  Arms: Short term memory assessment in patients with aphasia.
Diagnostic Test: Token Test — Evaluation of the severity of the aphasia in patients with aphasia.
  Arms: Short term memory assessment in patients with aphasia.
Diagnostic Test: Montreal cognitive assessment — Evaluation of cognitive dysfunction in the group of healthy volunteers.
  Arms: short term memory assessment in healthy volunteers

SUMMARY:
Background and aim

There is a growing awareness that people with aphasia (language problems) after a stroke often have difficulties with their short-term memory (STM). As a result, the explanation underlying aphasia has recently been seen as a language processing disorder, where multiple cognitive processes interact. To evaluate the cognitive processes underlying aphasia, there is a need for reliable and valid assessment tools. However, the quality of tests usually used to assess STM problems in aphasia patients is questioned because they are not specifically designed to be used in aphasia patients. This raises some concern, as impairments of STM can be predictive for the recovery and rehabilitation of aphasia patients. As an important exception, a recent study has developed a new English evaluation tool (i.e., The Temple Assessment of Language and (Verbal) Short-term Memory in Aphasia; TALSA) that examines language and STM aspects specifically developed for persons with aphasia.

However, the existence of a Dutch evaluation tool specifically designed to assess language and STM problems in people with aphasia after a stroke is lacking. Therefore, the aim of the current study is to develop a Dutch clinical version of the TALSA battery that may lead to better diagnosis and treatment of STM problems in persons with aphasia. The development of the test focuses on its clinical feasibility (e.g. test duration, difficulty of the items and response modality). Pilot testing of the Dutch STM assessment instrument in the clinical and healthy population is very important to adapt the test where necessary. In addition, the quality of the test should also be carefully evaluated.

Method

The first step towards the development of a Dutch STM assessment instrument is the careful selection of the most crucial subtests of the original TALSA battery. Not all subtests will be selected due to the long testing time of the TALSA battery, and as mentioned earlier, the Dutch STM assessment tool focuses on clinical feasibility of the test.

The second step is pilot testing the Dutch STM assessment instrument in persons with aphasia and healthy persons. Persons with aphasia will be recruited at the Stroke unit of Ghent University Hospital. All eligible patients will be asked to provide written informed consent to participate in this study. Three tests will be administered, namely the Oxford Cognitive Screen, the Token Test and the Dutch STM assessment tool. It is important that these tests are taken on the same day or on two consecutive days, depending on the circumstances (e.g. fatigue). The Token Test and Oxford Cognitive Screen provide a picture of the patient's cognitive profile. Throughout the process of pilot testing, the Dutch STM assessment tool will be adapted and improved where necessary. In order to verify or adjust the difficulty of the items, it is crucial that the STM assessment instrument is also tested on a small number of healthy control subjects (recruited via social media platforms).

DETAILED DESCRIPTION:
1. Introduction

   1.1. Background

   The literature has witnessed a steady increase in the number of studies investigating the role of short-term memory (STM) and working memory (WM) impairments in aphasia patients, which clearly shows that aphasia patients have impairments in verbal STM and WM. Throughout the years, views on the nature of aphasia have changed from the loss of linguistic representations (e.g., semantic and phonological representations) into impairments in the processing (i.e., access and retrieval) of language representations. Therefore, the emphasis of research has been refined in identifying the component operations of language processing, such as the mechanisms behind the access and retrieval of words or the temporal course of language processing. These operations rely on other cognitive functions, such as the STM.

   Psycholinguistic models describe the role of the STM in language as the maintenance of activation of linguistic representations over the time course of processing words. Particularly, the interactive activation model takes levels of linguistic representations (e.g., semantic, lexical and phonological) and its connections into account. Specifically, according to this influential model, word retrieval is mediated by interactive spreading activation that activates the target word and semantically or phonologically related words. Two important concepts (i.e., connection strength and decay rate) play an important role in spreading and maintaining activation over time in the semantic-lexical-phonological network. In aphasia, the impairments are thought to occur through deficits in linguistic representations, and moreover, through deficits in connection weight and decay rate (i.e., processing impairment). Errors occur if connection strength is weak (activation spreads too slowly) or if the decay rate is too rapid (representations are activated but decay too fast). Therefore, the interactive activation model can explain different patterns of word retrieval errors (i.e., semantical or phonological) in aphasia.

   In order to examine the role of the STM in language processing, there is an excessive need for reliable assessment tools. However, the psychometric properties of tests commonly used to assess STM problems in individuals with aphasia have been called into question. A common issue across these tests is that small standardized samples are used, which lead to validity and reliability problems of normative data. This raises some concerns since there is growing awareness that impairments in STM functions may be predictive of certain aspects of language function, recovery and rehabilitation in aphasia patients. Therefore, it is of crucial importance that STM assessment tools are reliable and valid in order to replicate, compare and further examine these findings.

   A recent study developed a new English assessment tool (i.e., The Temple Assessment of Language and (Verbal) Short-term Memory in Aphasia; TALSA) that evaluates language and verbal STM/WM abilities in individuals with poststroke aphasia in an interactive activation framework. In other words, to evaluate the nature of aphasia as a processing disorder. The TALSA battery is unique compared to other tests (e.g. Psycholinguistic assessments of language processing in aphasia (PALPA)) since it takes into account features related to temporal aspects of language processing and effects of memory load on production and comprehension of language. Therefore, the TALSA battery is a specific diagnostic assessment tool and is sensitive to language impairments at all levels of severity, including mild aphasia. The complete TALSA battery consists of three parts among which the last part involves verbal STM tasks. Note that the authors of the TALSA battery are still working on a clinical version that is not published yet.

   1.2. Rationale of the study

   To our knowledge, the existence of a Dutch assessment tool that examines verbal STM in individuals with poststroke aphasia is lacking. In other words, a Dutch STM test specifically developed for people with phatic disorders is not available. However, assessing non-linguistic influences in aphasia patients, such as the role of STM on language components, is of crucial importance as communication in everyday life fluctuates in processing time.

   Moreover, an overwhelming amount of STM measures (standardised and experimental) are used in aphasia research. However, diversity in STM tests makes it harder to compare discrepant findings and makes it more difficult for clinicians to select appropriate assessment tools. Furthermore, the validity and reliability of used STM tools are questioned in the aphasic population. Thus, the establishment of a Dutch verbal STM assessment tool is crucial to better comprehend the nature of aphasia as a processing disorder, and has the purpose to serve as a practical tool to help Dutch clinicians and speech pathologists diagnose STM deficits more specifically, which can lead to optimized speech therapy.

   1.3. Objective of the study

   The first aim of the present study is to develop a Dutch clinical verbal STM assessment tool, based on the third part of the TALSA battery, to assess STM deficits at all levels of severity. With this intention, the investigators hope to better comprehend the nature of aphasia and the impact of STM deficits which may ameliorate treatment techniques. Importantly, this test focuses on clinical use and administration, in which despite the patient's language problems, the test must be understandable and applicable (e.g., test duration and response modality).

   The second aim is to run a pilot test on the aphasic population and the healthy population. Running a pilot test will validate the stimuli and the wording of the tasks. Confounded items (e.g., ambiguous stimuli, poor wording) will be revised or eliminated if necessary.

   The third aim is to evaluate the verbal STM assessment tool with respect to important psychometric properties, as the methodological quality of a test affects the interpretation of the results.
2. Method

2.1. Study population

The investigators will include a maximum of 100 patients with aphasia in the acute to subacute phase after an ischemic or hemorrhagic stroke. The patients will be directly recruited in the Ghent University hospital at the Stroke unit. Furthermore, 20 healthy controls will be recruited via social media platforms. Healthy participants will be matched to the aphasic group for gender, age and education. All participants will voluntarily participate in this research project and sign an informed consent.

2.2. Verbal STM assessment tool development (first aim)

The first step towards the development of a Dutch clinical verbal STM assessment tool is to carefully select the most crucial verbal STM subtests of the original English TALSA battery. This is because the original TALSA battery is quite long and is not yet developed for administration in clinical settings. In particular, the Dutch verbal STM assessment tool will be based on the third part of the TALSA battery which involves verbal STM span tasks. The third part of the TALSA battery, moreover, evaluates phonological and semantic language representations by varying word characteristics of the items. Thus, the Dutch verbal STM assessment tool will consist of verbal STM span tasks with linguistic variations (phonological and semantic representations).

The stimuli in the original TALSA battery consist of pictures and recordings of words, nonwords, sentences, and sequences of words, nonwords, and digits. However, literally translating the TALSA test-battery is inappropriate because there is not a one-to-one match between words and syntactic structures across any two languages. In particular, it is important to take into account word characteristics, such as word frequency, syllables, imageability and age of acquisition, that influence the degree of success in word retrieval in aphasia. Therefore, the verbal STM assessment tool will rely on the same subset tasks of part 3 of the TALSA battery, but with the careful selection of new Dutch stimuli with respect to important word characteristics.

In the original TALSA battery, the authors took word frequency, syllables and imageability into account. However, research showed that age of acquisition (AoA) is also a crucial word characteristic in success of word retrieval in aphasia, thus AoA will be included during the stimuli selection procedure. In order to collect stimuli that meet these general word characteristics, word databases will be consulted, such as the Dutch Lexicon Project 2.

2.3. Pilot test (second aim)

Once the test-battery is developed, pilot testing will be of crucial importance in the clinical setting and healthy population to adapt and improve the test-battery where necessary.

Particularly in the clinical setting, patients with aphasia will be recruited according to the inclusion and exclusion criteria. Specifically, all patients who are eligible will be asked for informed consent to participate in this trial. Subsequently, the Oxford Cognitive screen, the Token Test and the Dutch verbal STM assessment tool will be administered.

The Token Test determines the severity of aphasia and investigates sentence comprehension. The Oxford Cognitive screen is a short cognitive screening tool that is administered in the acute phase of stroke. The outcomes on the Token Test and Oxford Cognitive Screen can serve as a support to interpret the results of the Dutch verbal STM assessment tool.

It is worth noting that the Dutch verbal STM assessment tool, the Token Test and the Oxford Cognitive screen will be administered over a time span of maximum two consecutive days depending on how fatigued the patient is during testing. The total test duration on patients is estimated to take approximately two hours. The total test duration on healthy controls is estimated to take approximately 1 hour. During administration of the Dutch verbal STM assessment tool, audio recordings will be made of the patient. In this way, it is possible to reevaluate misunderstandings during the scoring of the subtests.

In order to verify or adapt the difficulty of the items, it is critical that the Dutch verbal STM assessment tool will also be tested on healthy controls. Results of the original TALSA battery revealed that healthy controls performed near ceiling on most of the subtests. However, in some of the subtests (e.g., nonword span), healthy controls showed a similar results pattern as aphasia patients, which questions the contribution of those subtests.

To conclude, running a pilot test provides the opportunity to reevaluate items that stand out from the distribution of scores (e.g., sufficient number of healthy controls respond incorrectly to an item). Specifically, these items may be confounded and need to be eliminated or adapted (e.g., ambiguous stimuli).

2.4. Psychometric properties (third aim)

Reliability and validity are important psychometric properties. Reliability refers to the consistency, stability and accuracy of an assessment tool. Validity of a test refers to whether the assessment tool measures what it intends to measure.

* Internal consistency: To verify the reliability of the Dutch verbal STM assessment tool, the internal consistency of the test will be estimated using the split-half reliability procedure. In this way, the constancy of results across items within a subtest can be analyzed.
* Face validity: The TALSA battery is developed to approach aphasia as a processing disorder, supported by cognitive models of language processing. Therefore, the test battery focuses on component stages of word processing (e.g., semantic or phonological) and, moreover, with an emphasis on processes related to access, retrieval and short-term maintenance of language representations.
* Concurrent validity: The results of the Dutch verbal STM assessment tool will be compared with the results of the original TALSA battery to verify the concurrent validity. High correlations between the subtests of the original TALSA battery and Dutch verbal STM assessment tool suggest a good concurrent validity.

To conclude, throughout the process of pilot testing, the Dutch verbal STM assessment tool will be modified and improved where necessary and will be psychometrically evaluated (e.g., reliability, validity and item analysis).

ELIGIBILITY:
Inclusion Criteria aphasia patients:

* Aphasia after an initial ischemic or hemorrhagic stroke diagnosed by the speech pathologist and a screening instrument to evaluate aphasia (ScreeLing)
* Age 18-85 years
* Speak Dutch as a mother language
* Acute to subacute phase poststroke
* Imaging (CT/MRI) is available prior to inclusion
* Signed informed consent

Exclusion Criteria aphasia patients:

* There is a history of other diseases of the central nervous system causing non-stroke related speech-, language or cognitive disorder
* They present severe sensory impairment or other co-morbidities prohibiting administration of the assessment tool
* Excessive active alcohol or drug abuse
* Transient ischemic attack (i.e., TIA)

Inclusion Criteria healthy participants:

* Normal score (> 26) on the Montreal Cognitive Assessment (MOCA)
* Speak Dutch as a mother language

Exclusion Criteria aphasia patients:

* Have no history of stroke or other central nervous system diseases that affect speech, language or cognition
* Have no severe auditory or visual disorders

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2023-04-30 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
verbal short-term memory in poststroke aphasia | 2 hours
  assessment of verbal short-term memory in patients with poststroke aphasia: feasability, psychometric properties and normative data

CONTACTS AND LOCATIONS:
Locations (2):
- Belgium (2):
  - Ghent University Hospital, Ghent, East Flanders
  - University Hospital Ghent, Ghent

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] DE RENZI E, VIGNOLO LA. The token test: A sensitive test to detect receptive disturbances in aphasics. Brain. 1962 Dec;85:665-78. doi: 10.1093/brain/85.4.665. No abstract available. PMID 14026018
- [Background] Brysbaert M, Stevens M, Mandera P, Keuleers E. The impact of word prevalence on lexical decision times: Evidence from the Dutch Lexicon Project 2. J Exp Psychol Hum Percept Perform. 2016 Mar;42(3):441-58. doi: 10.1037/xhp0000159. Epub 2015 Oct 26. PMID 26501839
- [Background] Dell GS, O'Seaghdha PG. Stages of lexical access in language production. Cognition. 1992 Mar;42(1-3):287-314. doi: 10.1016/0010-0277(92)90046-k. PMID 1582160
- [Background] Dell GS, Schwartz MF, Martin N, Saffran EM, Gagnon DA. Lexical access in aphasic and nonaphasic speakers. Psychol Rev. 1997 Oct;104(4):801-38. doi: 10.1037/0033-295x.104.4.801. PMID 9337631
- [Background] Demeyere N, Riddoch MJ, Slavkova ED, Bickerton WL, Humphreys GW. The Oxford Cognitive Screen (OCS): validation of a stroke-specific short cognitive screening tool. Psychol Assess. 2015 Sep;27(3):883-94. doi: 10.1037/pas0000082. Epub 2015 Mar 2. PMID 25730165
- [Background] Harnish SM, Lundine JP. Nonverbal Working Memory as a Predictor of Anomia Treatment Success. Am J Speech Lang Pathol. 2015 Nov;24(4):S880-94. doi: 10.1044/2015_AJSLP-14-0153. PMID 26383918
- [Background] Ivanova MV, Hallowell B. A tutorial on aphasia test development in any language: Key substantive and psychometric considerations. Aphasiology. 2013 Jan 1;27(8):891-920. doi: 10.1080/02687038.2013.805728. PMID 23976813
- [Background] Lang CJ, Quitz A. Verbal and nonverbal memory impairment in aphasia. J Neurol. 2012 Aug;259(8):1655-61. doi: 10.1007/s00415-011-6394-1. Epub 2012 Jan 19. PMID 22258478
- [Background] Martin N, Gupta P. Exploring the relationship between word processing and verbal short-term memory: evidence from associations and dissociations. Cogn Neuropsychol. 2004 Mar 1;21(2):213-28. doi: 10.1080/02643290342000447. PMID 21038201
- [Background] Martin N, Minkina I, Kohen FP, Kalinyak-Fliszar M. Assessment of linguistic and verbal short-term memory components of language abilities in aphasia. J Neurolinguistics. 2018 Nov;48:199-225. doi: 10.1016/j.jneuroling.2018.02.006. PMID 30220790
- [Background] Mayer JF, Murray LL. Measuring working memory deficits in aphasia. J Commun Disord. 2012 Sep-Oct;45(5):325-39. doi: 10.1016/j.jcomdis.2012.06.002. Epub 2012 Jun 16. PMID 22771135
- [Background] Murray L, Salis C, Martin N, Dralle J. The use of standardised short-term and working memory tests in aphasia research: a systematic review. Neuropsychol Rehabil. 2018 Apr;28(3):309-351. doi: 10.1080/09602011.2016.1174718. Epub 2016 May 4. PMID 27143500
- [Background] Seniow J, Litwin M, Lesniak M. The relationship between non-linguistic cognitive deficits and language recovery in patients with aphasia. J Neurol Sci. 2009 Aug 15;283(1-2):91-4. doi: 10.1016/j.jns.2009.02.315. Epub 2009 Mar 6. PMID 19268973
- [Background] Bastiaanse, R, Wieling, M, Wolthuis, N. The role of frequency in the retrieval of nouns and verbs in aphasia. Aphasiology. 2016; 30(11): 1221-1239.
- [Background] Kay, J, Lesser, R, Coltheart, M. Psycholinguistic assessments of language processing in aphasia (PALPA): An introduction. Aphasiology. 1996; 10(2): 159-180.
- [Background] McNeil, MR, Pratt, SR. Defining aphasia: Some theoretical and clinical implications of operating from a formal definition. Aphasiology. 2001; 15(10-11): 901-911.
- [Background] Murray, LL. Direct and indirect treatment approaches for addressing short-term or working memory deficits in aphasia. Aphasiology. 2012; 26(3-4): 317-337.
- [Background] Dell GS, Martin N, Schwartz MF. A Case-Series Test of the Interactive Two-step Model of Lexical Access: Predicting Word Repetition from Picture Naming. J Mem Lang. 2007 May 1;56(4):490-520. doi: 10.1016/j.jml.2006.05.007. PMID 21085621